CLINICAL TRIAL: NCT00163384
Title: A Comparative Study of Inhaled Ciclesonide 160 mcg/Day vs Budesonide 400 mcg/Day in Patients With Asthma
Brief Title: Effectiveness of Ciclesonide Versus Budesonide in Patients With Asthma (18 to 75 y) (BY9010/M1-136)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-136
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Budesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
This trial will compare the effectiveness of one dose of ciclesonide against one dose of budesonide in patients with asthma.

The aim of the present trial is to compare the efficacy of ciclesonide versus budesonide on pulmonary function, symptoms and use of rescue medication in patients with asthma. The onset of action and the safety and tolerability of ciclesonide in comparison to budesonide will also be investigated.

ELIGIBILITY:
Main Inclusion Criteria:

* During the last 4 weeks prior to baseline, treatment with an inhaled steroid (dosage: up to 250 mcg fluticasone propionate or equivalent)
* FEV1 80 - 105% of predicted
* Healthy with the exception of asthma
* Written informed consent has been obtained
* Outpatients
* Patients who have a history of persistent bronchial asthma for at least 6 months

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Concomitant COPD (chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* An asthma exacerbation or an infection of the lower airways prior to entry into the baseline period
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception
* Patient is current smoker with 10 or more pack-years
* Patient is ex-smoker with 10 or more pack-years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2004-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
FEV1 absolute values.

SECONDARY OUTCOMES:
FEV1 as percent of predicted
FVC
PEF absolute values
morning and evening PEF from diary
diurnal PEF fluctuation
asthma symptom score from diary
use of rescue medication from diary
number of symptom free- and rescue medication free days
dropout rate due to asthma exacerbations
time until first asthma exacerbation
number of days with asthma control
onset of effect
subgroup analysis for ex/current smokers and non-smokers
AQLQ(S).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (10):
- South Korea (10):
  - Altana Pharma/Nycomed, Busan
  - Altana Pharma/Nycomed, Daegu
  - Altana Pharma/Nycomed, Daejeon
  - Altana Pharma/Nycomed, Gangwon-do
  - Altana Pharma/Nycomed, Gwangju
  - Altana Pharma/Nycomed, Gyeonggi-do
  - Altana Pharma/Nycomed, Jeonju
  - Altana Pharma/Nycomed, Jungbuk
  - Altana Pharma/Nycomed, Jungnam
  - Altana Pharma/Nycomed, Seoul

REFERENCES:
- See also: BY9010-M1-136-RDS-2006-12-03.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4521&filename=BY9010-M1-136-RDS-2006-12-03.pdf